CLINICAL TRIAL: NCT06096441
Title: Clinical and Molecular Characterization of Facioscapulohumeral Muscular Dystrophy (FSHD)
Brief Title: FSHD Molecular Characterization
Status: Terminated | Type: Observational
Why Stopped: This study was closed due to inability to to recruit.
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Kevin Flanigan, Director, Center for Gene Therapy, Professor of Pediatrics and Neurology, Nationwide Children's Hospital
Other Study IDs: STUDY00001521
Record Dates: First submitted 2023-09-12; First posted 2023-10-23 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Facio-Scapulo-Humeral Dystrophy
Keywords: FSHD
MeSH Terms: conditions — Muscular Dystrophy, Facioscapulohumeral

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Collecting blood products (plasma and serum for RNA and DNA) and muscle biopsies.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
To characterize the clinical and molecular phenotype of FSHD.

DETAILED DESCRIPTION:
The purpose of this study is to validate alterations in therapeutically relevant biomarkers in muscle tissue from FSHD patients. These biomarkers are responsive to the upregulation of the DUX4 gene and protein, which is the fundamental molecular defect in FSHD. In anticipation of a future clinical trial, the Investigators intend to assess the correlation between the expression of these relevant biomarkers and clinical functional measures. The Investigators will also explore the utility of muscle MRI in identifying regions of muscle suitable for sampling for relevant biomarkers, as MRI-related signal changes have been proposed as an anatomic marker of early FSHD pathology.

ELIGIBILITY:
Inclusion Criteria:

* 13 years or older
* Genetically proven FSHD1 or FSHD2 as determined by the investigators

Exclusion Criteria:

* Inability to complete an MRI scan (Adults only).
* Other medical or cognitive issues that, in the opinion of the examiner, preclude accurate functional assessment.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects 13 years or older with facioscapulohumeral muscular dystrophy (FSHD).
Sampling Method: Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2021-03-05 (Actual); Primary Completion 2025-09-09 (Actual); Study Completion 2025-09-09 (Actual)

PRIMARY OUTCOMES:
Validation of Biomarkers | Through study completed, anticipated to be 4 years.
  To validate alterations in therapeutically relevant biomarkers in muscle tissue from FSHD participants. Each participant will provide data at a single timepoint. The data in totality will be reviewed upon study completion.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Flanigan, MD, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- The Abigail Wexner Research Institute at Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided
We will be willing to share de-identified data following the execution of a Data Use Agreement.

REFERENCES:
- [Background] Amini Chermahini G, Rashnonejad A, Harper SQ. RNAscope in situ hybridization-based method for detecting DUX4 RNA expression in vitro. RNA. 2019 Sep;25(9):1211-1217. doi: 10.1261/rna.070177.118. Epub 2019 Jun 17. PMID 31209064
- [Background] Jones TI, Chen JC, Rahimov F, Homma S, Arashiro P, Beermann ML, King OD, Miller JB, Kunkel LM, Emerson CP Jr, Wagner KR, Jones PL. Facioscapulohumeral muscular dystrophy family studies of DUX4 expression: evidence for disease modifiers and a quantitative model of pathogenesis. Hum Mol Genet. 2012 Oct 15;21(20):4419-30. doi: 10.1093/hmg/dds284. Epub 2012 Jul 13. PMID 22798623
- [Background] Snider L, Asawachaicharn A, Tyler AE, Geng LN, Petek LM, Maves L, Miller DG, Lemmers RJ, Winokur ST, Tawil R, van der Maarel SM, Filippova GN, Tapscott SJ. RNA transcripts, miRNA-sized fragments and proteins produced from D4Z4 units: new candidates for the pathophysiology of facioscapulohumeral dystrophy. Hum Mol Genet. 2009 Jul 1;18(13):2414-30. doi: 10.1093/hmg/ddp180. Epub 2009 Apr 9. PMID 19359275
- [Background] Wang LH, Friedman SD, Shaw D, Snider L, Wong CJ, Budech CB, Poliachik SL, Gove NE, Lewis LM, Campbell AE, Lemmers RJFL, Maarel SM, Tapscott SJ, Tawil RN. MRI-informed muscle biopsies correlate MRI with pathology and DUX4 target gene expression in FSHD. Hum Mol Genet. 2019 Feb 1;28(3):476-486. doi: 10.1093/hmg/ddy364. PMID 30312408
- [Background] Yao Z, Snider L, Balog J, Lemmers RJ, Van Der Maarel SM, Tawil R, Tapscott SJ. DUX4-induced gene expression is the major molecular signature in FSHD skeletal muscle. Hum Mol Genet. 2014 Oct 15;23(20):5342-52. doi: 10.1093/hmg/ddu251. Epub 2014 May 26. PMID 24861551